CLINICAL TRIAL: NCT03263715
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy of Tocilizumab as a Remission-Induction and Glucocorticoid-Sparing Regimen in Subjects With New-Onset Polymyalgia Rheumatica (PMR- SPARE)
Brief Title: A Study to Evaluate the Efficacy of Tocilizumab as a Remission-Induction and Glucocorticoid-Sparing Regimen in Subjects With New-Onset Polymyalgia Rheumatica (PMR- SPARE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Daniel Aletaha, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PMR-SPARE; 2016-004990-42 (EudraCT Number)
Record Dates: First submitted 2017-08-17; First posted 2017-08-28 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Polymyalgia Rheumatica
Keywords: Polymyalgia Rheumatica; Tocilizumab; Glucocorticoid; Glucocorticoid-Sparing
MeSH Terms: conditions — Polymyalgia Rheumatica | interventions — tocilizumab; Glucocorticoids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tocilizumab (Experimental): Tocilizumab-based regimen (Tocilizumab Prefilled Syringe [Actemra] 162 mg s.c. administered weekly) on top of rapidly tapered Glucocorticoid [Glucocorticoids]
  Interventions: Drug: Tocilizumab Prefilled Syringe [Actemra]; Drug: Glucocorticoids
- Placebo (Placebo Comparator): Placebo [Placebos] and rapidly tapered Glucocorticoid [Glucocorticoids] treatment
  Interventions: Drug: Placebos; Drug: Glucocorticoids

INTERVENTIONS:
Drug: Tocilizumab Prefilled Syringe [Actemra] — Weekly administration of Tocilizumab 162 mg subcutaneous from Baseline to Week 16.
  Other Names: Actemra
  Arms: Tocilizumab
Drug: Placebos — Weekly administration of Placebo subcutaneous from Baseline to Week 16.
  Arms: Placebo
Drug: Glucocorticoids — Rapidly tapered Glucocorticoid treatment. 20 mg/day of prednisone at randomization and a pre-specified taper regimen will be followed over 11 weeks: Week 0: 20 mg Week 1: 17,5 mg Week 2: 15 mg Week 3: 12,5 mg Week 4: 10 mg Week 5: 9 mg Week 6: 7 mg Week 7: 5 mg Week 8: 4 mg Week 9: 2 mg Week 10: 1 mg Week 11: 0 mg

SUMMARY:
The purpose of this study is to assess the efficacy of a tocilizumab-based regimen compared with placebo on top of rapidly tapered glucocorticoid treatment in a double- blind, controlled fashion, focussing on glucocorticoid-free remission of disease.

DETAILED DESCRIPTION:
Background. Polymyalgia rheumatica is an inflammatory rheumatic disease of the elderly, with a usually rapid response to intermediate-doses of glucocorticoids (GCs). In many patients, relapses occur upon its dose reduction or cessation. Given the patients' age and the adverse event profile of GCs, steroid- free remission is the most desired target in patients with PMR, but typical GC sparing agents are often insufficient. Case series and small open studies suggested an excellent effectiveness of tocilizumab, an inhibitor of the Interleukin 6-receptor.

Objective. To assess the efficacy and safety of a tocilizumab-based regimen compared with placebo on top of rapidly tapered GC treatment in a double-blind, controlled fashion, focussing on GC-free remission of disease.

Methods. In this double-blind, parallel group study, 32 patients with PMR will be recruited from three rheumatology centres and will be randomised in a 1:1 ratio to tocilizumab or placebo over the course of 16 weeks, accompanied by a rapid tapering GC scheme over 11 weeks in both arms. The primary endpoint is GC-free remission at week 16, and follow-up will be performed until week 24 for safety and sustained efficacy. Patients will receive either the subcutaneous preparation of 162 mg tocilizumab weekly or matching placebo injections.

Expected Results. In case of a positive result of this study, the benefits for patients with new-onset PMR will manifest in a reduction of the burden of GC intake in this elderly population with increased risk of GC-related adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PMR as confirmed by the investigator at screening and at baseline, fulfilment (also in retrospect) of the provisional 2012 ACR- EULAR classification criteria
* Diagnosis of PMR established at, or up to 2 weeks before the screening visit
* GC naïve or on GC treatment for a maximum of 2 weeks at screening with an initial dose between 12.5 and 25mg/day prednisone
* Willing and able to receive oral prednisone 20mg/day at randomization and to follow a pre-specified tapering regimen
* Willing to receive treatment for prevention of GC-induced bone loss
* No evidence of active infection with Mycobacterium tuberculosis (screening performed according to national guidelines) and willing to take TB prophylaxis in case of evidence of latent TB
* Willing and being able to understand and follow the study procedures
* Male and female subjects agreeing to conduct efficient contraception (unless they have no childbearing potential)
* Written informed consent.
* Female and Male subjects from 18 years old and higher

Exclusion Criteria:

* Evidence of GCA (cranial or large vessel) as indicated by unequivocal clinical symptoms (except PMR), imaging and/or biopsy results. Routine screening of eligible PMR patients for GCA with imaging methods or temporal artery biopsy is not recommended
* GC treatment of PMR >2 weeks
* Conditions other than PMR requiring continuous or intermittent treatment with oral or parenteral GCs or parenteral administration of GCs, unless the last exposure to GCs was >1 months before screening
* Other inflammatory rheumatic diseases (e.g. rheumatoid arthritis)
* Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following randomization
* Treatment with any investigational agent within 4 weeks (or 5 half-lives of the investigational drug, whichever is longer) of screening
* Previous treatment with any cell-depleting therapies, including investigational agents or approved therapies, some examples include: CAMPATH, anti-CD4, anti-CD5, anti-CD3, anti-CD19 and anti-CD20
* Treatment with intravenous gamma globulin, plasmapheresis or Prosorba column within 6 months of baseline
* Immunization with a live/attenuated vaccine within 4 weeks prior to baseline
* Previous treatment with Tocilizumab (an exception to this criterion may be granted for single dose exposure upon application to the sponsor on a case-by-case basis)
* Any previous treatment with alkylating agents such as chlorambucil, or with total lymphoid irradiation
* History of severe allergic or anaphylactic reactions to human, humanized or murine monoclonal antibodies
* Evidence of serious uncontrolled concomitant cardiovascular, nervous system, pulmonary (including obstructive pulmonary disease), renal, hepatic, endocrine (include uncontrolled diabetes mellitus) or gastrointestinal disease (including complicated diverticulitis, ulcerative colitis, or Crohn ́s disease)
* Diagnosis of liver disease or elevated hepatic enzymes, as defined by ALT, AST, or both > 1.5 x the upper limit of age-determined normal (ULN) or total bilirubin > ULN
* Serum creatinine > 1.6 mg/dL (141 μmol/L) in female patients and > 1.9 mg/dL (168 μmol/L) in male patients. Patients with serum creatinine values exceeding limits may be eligible for the study, if their estimated glomerular filtration rates (GFR) are > 30
* Total Bilirubin > ULN
* Any history of recent serious bacterial, viral, fungal, or other opportunistic infections
* Have serologic evidence of current or past HIV, Hepatitis B, or Hepatitis C
* Positive QuantiFERON TB test, history of Tuberculosis, or active Tuberculosis-infection, without at least 4 weeks of adequate therapy for Tuberculosis
* Active infection with EBV as defined by EBV viral load > 10,000 copies per mL of whole blood
* Any of the following hematologic abnormalities, confirmed by repeat tests:

  1. White blood count < 3,000/μL or > 14,000/μL;
  2. Lymphocyte count < 500/ μL;
  3. Platelet count < 100,000/μL;
  4. Hemoglobin < 8.0 g/dL; or
  5. Neutrophil count < 2,000 cells/μL
* Any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening
* Primary or secondary immunodeficiency (history of or currently active) unless related to primary disease under investigation
* Any medical or psychological condition that in the opinion of the Principal Investigator would interfere with safe completion of the trial
* History of other malignancy within 5 years prior to screening, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or Stage I uterine cancer
* Pregnant women or nursing (breast feeding) mothers
* Patients with reproductive potential not willing to use an effective method of contraception
* History of alcohol, drug or chemical abuse within 1 year prior to screening
* Neuropathies or other conditions that might interfere with pain evaluation unless related to primary disease under investigation
* Patients with lack of peripheral venous access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-11-24 (Actual); Primary Completion 2020-06-02 (Actual); Study Completion 2020-06-02 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects in GC free remission at week 16 | Week 16
  Proportion of subjects in GC free remission at week 16

SECONDARY OUTCOMES:
Cumulative prednisone doses at weeks 12, 16 and 24 | Week 12, 16, 24
  Cumulative prednisone doses at weeks 12, 16 and 24
Number of flares per patient at weeks 12, 16 and 24 | Week 12, 16, 24
  Number of flares per patient at weeks 12, 16 and 24
Time to first and second flare | 24 Weeks
  Time to first and second flare
Patient reported outcomes including SF-36 | 24 Weeks
  Patient reported outcomes including SF-36
Patient reported outcomes including FACIT-Fatigue | 24 Weeks
  Patient reported outcomes including FACIT-Fatigue
Patient reported outcomes including HAQ | 24 Weeks
  Patient reported outcomes including HAQ
Patient reported outcomes including Patient Global Assessment of disease (PGA) | 24 Weeks
  Patient reported outcomes including Patient Global Assessment of disease (PGA)
Patient reported outcomes including Patient Assessment of pain | 24 Weeks
  Patient reported outcomes including Patient Assessment of pain
Investigator reported outcomes including Evaluator Global Assessment of disease activity (EGA) | 24 Weeks
  Investigator reported outcomes including Evaluator Global Assessment of disease activity (EGA)
Investigator reported outcomes including Duration and severity of Morning Stiffness | 24 Weeks
  Investigator reported outcomes including Duration and severity of Morning Stiffness
Investigator reported outcomes including Elevation of upper limbs | 24 Weeks
  Investigator reported outcomes including Elevation of upper limbs
Occurrence of adverse events and serious adverse events, incidence of GC related adverse events, changes in vital signs, haematology and clinical chemistry parameters | 24 Weeks
  Occurrence of adverse events and serious adverse events, incidence of GC related adverse events, changes in vital signs, haematology and clinical chemistry parameters
Proportion of subjects with increased ESR (>20mm/h) and CRP levels (> 5mg/L) at week 24 | Week 24
  Proportion of subjects with increased ESR (>20mm/h) and CRP levels (> 5mg/L) at week 24

CONTACTS AND LOCATIONS:
Locations (3):
- Austria (3):
  - Medizinische Universität Graz, Klinische Abteilung für Rheumatologie und Immunologie, Graz
  - Allgemeines Krankenhaus der Stadt Wien, Vienna
  - Krankenhaus Hietzing, 2. Medizinische Abteilung, Vienna

REFERENCES:
- [Derived] Bonelli M, Radner H, Kerschbaumer A, Mrak D, Durechova M, Stieger J, Husic R, Mandl P, Smolen JS, Dejaco C, Aletaha D. Tocilizumab in patients with new onset polymyalgia rheumatica (PMR-SPARE): a phase 2/3 randomised controlled trial. Ann Rheum Dis. 2022 Jun;81(6):838-844. doi: 10.1136/annrheumdis-2021-221126. Epub 2022 Feb 24. PMID 35210264